CLINICAL TRIAL: NCT00844584
Title: Clinical Study of Radiofrequency Ablation of Atrial Fibrillation Under Totally Thoracoscope
Brief Title: Radiofrequency Ablation of Atrial Fibrillation Under Totally Thoracoscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Jin Zhenxiao, Xijing Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: xinzangwaike0001
Record Dates: First submitted 2009-01-14; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; radiofrequency; totally thoracoscope; epicardial
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ablation (Other): patients with atrial fibrillation underwent radiofrequency ablation with totally thoracoscope.
  Interventions: Procedure: epicardial radiofrequency ablation

INTERVENTIONS:
Procedure: epicardial radiofrequency ablation — epicardial radiofrequency ablation to treat atrial fibrillation under totally thoracoscope
  Other Names: radiofrequency ablation

SUMMARY:
Atrial fibrillation (AF) is a common supraventricular arrhythmia, the incidence of which increases with age. The aim of treatment of atrial fibrillation is to restore sinus rhythm and return the heart to atrioventricular synchrony, avoiding the risk of thromboembolism. The fact that pharmacological therapy of AF is at best 50% effective has led to a search for surgical approaches over the last 20 years.

Maze procedure was a classic method to treat AF. However, it is such a complex procedure that very few surgeons have adopted it. A few minimally invasive procedures to create transmural lesions which mimic MAZE procedure have been introduced. One of the mostly favored methods is catheter-based radiofrequency ablation, another one is video assisted epicardial radiofrequency ablation through small thoracic incisions in operating room.

Recently, we invented an epicardial radiofrequency ablation method under totally thoracoscope, which further minimized the surgery trauma and increased the cosmetic effect.

ELIGIBILITY:
Inclusion Criteria:

* Any patients with atrial fibrillation

Exclusion Criteria:

* Patients with hemostasis defects
* patients can not endure general anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Electrocardiography | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dinghua Yi, MD, Study Director — Xijing Hospital
Locations (1):
- Institute of Cardiovascular Surgery, Xijing Hospital, Xi'an, Shannxi, China